CLINICAL TRIAL: NCT01320436
Title: Randomized, Double-blind, Placebo-controlled Study to Evaluated the Efficacy of Combining Curcumin+5ASA Medication Versus 5ASA Medication Alone on Active Mild to Moderate Ulcerative Colitis Patients
Brief Title: Curcumin + Aminosalicylic Acid (5ASA) Versus 5ASA Alone in the Treatment of Mild to Moderate Ulcerative Colitis
Acronym: 5ASA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Alon Lang, MD, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHEBA-10-8356-AL-CTIL
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; Curcumin
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Curcumin; Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatments arm (Active Comparator): Patients allocated for this arm will receive 5ASA medication (as advised by their treating physician) + 3 capsules (total of 820 mg each,containing 500 mg curcumin ) curcumin twice daily after meals.
  Interventions: Dietary Supplement: Curcumin; Drug: 5-aminosalicylic acid
- Control arm (Placebo Comparator): Patients allocated to this arm will receive 5ASA medication (as advised by their treating physician) + 3 capsules (820gr each) of placebo twice a day after meals.
  Interventions: Drug: 5-aminosalicylic acid

INTERVENTIONS:
Dietary Supplement: Curcumin — 3 capsules (820 mg containig 500 mg curcumin each) twice daily.
  Arms: Treatments arm
Drug: 5-aminosalicylic acid — The dosage of 5ASA medication will be the maximum dosage given in this group of patients according to clinical guidelines (4gr' per os + topical 1gr mesalamine
  Other Names: Pentasa, Asacol, Rafasal, Mesalamine.

SUMMARY:
Ulcerative colitis (UC) is a chronic inflammatory disease resulting in increased morbidity in patients. The current standard treatment for mild to moderate UC (MTMUC) includes 5-aminosalicylic compounds (5ASA) such as olsalazine and mesalamine, yet some patients continue to experience disease symptoms and flare-ups. These patients require higher dosages of 5ASA medications and in many cases escalate to steroid and/or immunosuppressant therapy which comprises higher risk of hazardous side effects.

Curcumin, an active ingredient of the Indian herb Rhizoma Curcuma Longa, has been extensively studied in the context of inflammatory diseases. In humans, a controlled study using curcumin as an adjusted therapy to 5ASA medication has shown it to be superior to placebo in maintaining remission in MTMUC patients . A small, preliminary open label study has also shown efficacy in reducing disease symptoms and inflammatory markers in this group of patients .

This data provides bases for investigating an integrative approach to optimize the current standard treatment in MTMUC patients. We speculate that using a combined therapy of 5ASA medication and curcumin could benefit this subgroup of patients and reduce morbidity and perhaps need for escalating pharmacological intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of UC as confirmed by endoscopic or histologic criteria as established by RomeIII
* Disease activity score of >5 and ≤13 according to the Simple clinical colitis activity index (SCCAI)
* Patient on stable 5 ASA medication dose for at least 4 weeks prior to inclusion
* Patients who receive immunosuppressant or biological therapy (azathioprine, 6-mercaptopurine, infliximab or methotrexate) must be on stable dose for at least 3 months prior to inclusion
* Patients who receive topical therapy (5ASA or steroidal), must be on stable dose for a least 2 weeks prior to inclusion
* Patient had hemoglobin of >10 g/dl.
* Able and willing to give written consent

Exclusion Criteria:

* Patient with renal or liver disease, sever cardiovascular disease, chronic pancreatitis, diabetes mellitus or gallstone.
* Patient with laboratory abnormalities indicating anemia (hemoglobin <10), leucopenia, thrombocytopenia, abnormal coagulation.
* Patient with infection, sepsis or pneumonia.
* Pregnant or nursing women.
* Unable or unwilling to receive CURCUMIN therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-07; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The percentage of patients who achieve clinical remission compared between the two study arms. | 4 weeks
  The percentage of patients who achieve clinical remission compared between the two study arms at week 4 after induction of therapy. Clinical remission is defined as score of ≤2 in the Simple Clinical Colitis Activity Index (SCCAI) .

SECONDARY OUTCOMES:
Time to response | 4 weeks
  Time to response (TTR) compared between study and control groups. Response is defined as remission or significant improvement. TTR is defined by number of days to achieve clinical response.
significant improvement | 4 weeks
  Percentage of patients that show significant improvement (drop of ≥3 points in SCCAI) compared between the two study arms at week 4 after induction of therapy.
serologic markers | 4 weeks
  Improvement in serologic parameters according to Seo index
Percentage of patient on corticosteroids or anti TNF treatment | 4 weeks
improvement in endoscopic score | 4 weeks
  Improvement in endoscopic score compared to inclusion day (in subgroup of patients)
Improvement in IBD questionnaire (IBDQ). | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alon Lang, MD, Principal Investigator — Sheba Medical Center; Nir Salomon, C.Ac, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Derived] Lang A, Salomon N, Wu JC, Kopylov U, Lahat A, Har-Noy O, Ching JY, Cheong PK, Avidan B, Gamus D, Kaimakliotis I, Eliakim R, Ng SC, Ben-Horin S. Curcumin in Combination With Mesalamine Induces Remission in Patients With Mild-to-Moderate Ulcerative Colitis in a Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2015 Aug;13(8):1444-9.e1. doi: 10.1016/j.cgh.2015.02.019. Epub 2015 Feb 24. PMID 25724700